CLINICAL TRIAL: NCT00848419
Title: A Prospective Randomized Comparison of Fentanyl, Methadone and Morphine for Epidural Analgesia in an Experimental Pain Model
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Exp pain 1-ginosar-HMO-CTIL
Record Dates: First submitted 2009-02-19; First posted 2009-02-20 (Estimated); Last update posted 2019-09-12 (Actual); Status verified 2009-02

CONDITIONS: Pain
Keywords: Epidural; Analgesia; Methadone; Morphine; Pharmacokinetic-pharmacodynamic; Experimental pain - analgesic response
MeSH Terms: conditions — Pain; Agnosia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Methadone (Active Comparator): Epidural methadone bolus 4mg
  Interventions: Drug: Epidural administration of bolus
- Morphine (Active Comparator): Epidural morphine 4mg bolus
  Interventions: Drug: Epidural administration of bolus
- Fentanyl (Active Comparator): Epidural fentanyl 200 microgram bolus
  Interventions: Drug: Epidural administration of bolus
- Saline (Placebo Comparator): Epidural saline bolus
  Interventions: Drug: Epidural administration of bolus

INTERVENTIONS:
Drug: Epidural administration of bolus

SUMMARY:
The aims of this study are to provide pharmacokinetic-pharmacodynamic data to quantify the analgesic and side effect profiles of epidural methadone, fentanyl and morphine. The investigators will compare the analgesic effect at three dermatomes to assess the rostral spread of drug, the investigators will assess plasma levels to assess the systemic redistribution of drug and the investigators will assess surrogate markers of central opiate effects (nasal capnography and pupilometry). The investigators hypothesize that due to the long-duration of action of methadone, and its intermediate lipophilicity, that methadone will provide a predominantly segmental analgesia of long duration of action, with low rostral spread and low direct central depressant effects (including respiratory depression).

ELIGIBILITY:
Inclusion Criteria:

* Patients (men and women) scheduled for extracorporeal shock wave lithotrypsy (for nephrolithiasis) under regional anesthesia.

Exclusion Criteria:

* Inability to understand consent form; poor communication Refusal to sign consent form Contraindication to regional anesthesia Chronic opioid administration ASA classification 3 or greater Age < 18 or > 70

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-04; Primary Completion 2009-12 (Estimated); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Change in heat pain tolerance from baseline (using QST Medoc) | At intervals: 30, 60, 90, 120, 180, 240, 300, 360, 410 min following drug and 24 hours following drug.

SECONDARY OUTCOMES:
Change in electrical pain tolerance from baseline | At same time intervals as primary outcome
Plasma concentration of methadone, fentanyl, morphine (and metabolites) | At each of the time intervals as for primary endpoint
Pupilometry | At each of the time intervals as primary endpoint
Respiratory rate and arterial CO2 tension | At each of the time intervals as primary endpoint